CLINICAL TRIAL: NCT06977945
Title: Clinical Application of FL-091 Radionuclide Imaging in Diagnosis and Staging of Malignant Tumors
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: XLan-0505
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Malignant Tumors With Positive NTSR1 Expression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1
  Interventions: Diagnostic Test: Specific positron imaging agents targeting NTRS-1(FL-091)

INTERVENTIONS:
Diagnostic Test: Specific positron imaging agents targeting NTRS-1(FL-091) — This study is diagnostic. Oncologists screen patients with malignant tumors such as head and neck cancer, colorectal cancer, and pancreatic adenocarcinoma who are clinically suspected or confirmed; investigators talk to patients who meet the inclusion criteria, explain the study purpose and study process, sign informed consent forms, and patients can complete 68Ga-FL-091PET imaging and 111In-FL-091SPECT imaging respectively in outpatient or inpatient periods. General information, clinical data, blood routine, urine routine, liver and kidney function and other biochemical indicators, electrocardiogram, radionuclide imaging results and other imaging data of the patients participating in the study were collected and compared with histopathology to evaluate the value of both imaging in the diagnosis of head and neck cancer, colorectal cancer, and pancreatic adenocarcinoma.

SUMMARY:
Malignant tumors pose a serious threat to human health, and early diagnosis and early treatment are crucial to improving the patient's prognosis. Nuclear medicine imaging technology injects radioisotope labeled molecules (such as monoclonal antibodies and peptides) into the body to identify and bind specific targets of different tumor cells, thereby achieving accurate early diagnosis of different tumors. Neurotensin receptor 1 (NTSR1) is overexpressed in many malignant tumors such as colon cancer, pancreatic cancer, gastric cancer, head and neck cancer, and is closely related to tumor occurrence, development and prognosis. At the same time, NTSR1 is low expressed in surrounding normal tissues, so NTSR1 is an excellent target for the diagnosis and diagnosis of the above-mentioned series of malignant tumors. Probes targeting NTSR1 have been gradually explored. FL-091 is a new NTSR1-targeted radionuclide conjugated drug (RDC) that has high affinity and specificity for NTSR1 in previous preclinical studies. Compared with conventional NTSR1 inhibitors, FL-091 has the following potential advantages: ① Potential for radiotherapy: FL-091 can combine with radioactive isotopes such as 177Lu or 225Ac to directly deliver radioactive energy to tumor cells. This radiation therapy can produce cytotoxicity in a local area, killing tumor cells while causing less damage to surrounding healthy tissues;② Selectivity and specificity: Since FL-091 is designed based on the high affinity of NTSR1, it can more selectively target tumor cells that express NTSR1. This high degree of specificity can reduce the impact on normal cells and increase the accuracy of imaging and treatment.③ Biodistribution and rapid clearance: FL-091 demonstrated optimized biodistribution characteristics, such as higher tumor uptake rates and faster clearance of normal tissues. This means it can effectively deliver radioactive material to tumor tissue while reducing radiation exposure to healthy tissue. Based on the above advantages, FL-091 labeled with imaging nuclide or therapeutic nuclide is expected to be used for precise imaging and treatment of targeted NTSR1, bringing new diagnosis and treatment methods to patients.

In this project, it is planned to use 68Ga and 111In to label FL-091 respectively for PET or SPECT imaging to initially evaluate the biodistribution of the probe in the human body, and diagnose and stage various malignant tumors including head and neck cancer, colorectal cancer and pancreatic adenocarcinoma. We will discuss the detection performance of 68Ga-FL-091 and 111In-FL-091 on malignant tumors, and lay the foundation for future use of therapeutic nuclide labeled FL-091 for nuclide targeted internal irradiation treatment of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all enrollment criteria to be eligible to participate in the study:

1. The subject or his/her legal representative is able to sign and date the informed consent form;
2. A commitment to comply with the research procedures and to cooperate in the implementation of the full research process;
3. Adult patients or healthy volunteers (aged 18 or above) of either sex;
4. Patients with clinically suspected or confirmed malignant tumors such as head and neck cancer, colorectal cancer, or pancreatic cancer (supporting evidence includes serum-related tumor markers, imaging data such as ultrasound, CT, MRI, etc., and histological pathology examination, etc.) and in good general condition;
5. Consistent with the results of specific laboratory tests;
6. Females of childbearing potential who have been using contraception for at least one month prior to screening and who are committed to using contraception for the entire study period and until a specified time after the end of the study；
7. Other set entry criteria.

Exclusion Criteria:

All subjects who meet any of the exclusion criteria baseline will be excluded from the study:

1. Those who are unable to complete a PET/MR or PET/CT examination (including inability to lie down, claustrophobia, radiophobia, etc.);
2. Having other comorbidities;
3. Patients with known hypersensitivity to FL-091 fragment developers or synthetic excipients; fasting blood glucose level greater than 11.0 mmol/L prior to 18F-FDG injection；
4. Have a history of comorbid drug use;
5. Patients considered by the investigator to have poor compliance;
6. Patients during pregnancy or lactation;
7. Persons with other factors that make participation in this test inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected or confirmed malignant tumors such as head and neck cancer, colorectal cancer, or pancreatic cancer (supporting evidence includes serum-related tumor markers, imaging data such as ultrasound, CT, MRI, etc., and histological pathology examination, etc.) and in good general condition.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting NTSR-1 nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Pathological sections of tumour tissue | 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its NTSR-1 expression

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital,China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided